CLINICAL TRIAL: NCT04661722
Title: Comparison of Prognostic Performance of TIMI, GRACE, HEART and HEARTSIL SCORES in Patients Admitted to the Emergency Department With Chest Pain
Brief Title: A Comparison of the TIMI, GRACE, HEART and HEARTSIL Scores
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Nazire B Akilli,MD, associate professor, Konya Meram State Hospital
Other Study IDs: Konya city hospital
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2020-12

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Chest pain is one of the most common reasons for emergency admission. Chest pain can be caused by many cardiac and noncardiac causes. Acute Coronary Syndrome (ACS) is one of the most im-portant of these etiologies. ACS has a high mortality rate, but with early diagnosis and related inter-ventions, a high rate of prognosis can be improved. Therefore, early recognition of AKS is impor-tant. However, the challenge in emergency services is not only to identify patients with high risk for ACS. Early detection of low-risk patients is also important for emergency room management. These patients should be discharged quickly with minimal examination and treatment. The follow-up of these patients with the acceptance of ACS brings along unnecessary examinations and treatments. This leads to an increase in healthcare costs and an increase in crowd in emergency services and hospitals.

Evaluation of chest pain in the emergency room and early detection of life-threatening conditions such as ACS present many difficulties for clinicians. For this reason, clinicians use some scoring systems that determine the risk stratification of patients and the probability of having acute coronary syndrome. Heart score is one of the scores developed for this purpose. However vital signs are not included in calculating the heart score. Therefore, the investigators considered to include the shock index calcula-ted by systolic blood pressure and pulse in this scoring system. In addition, the investigators have included a very valuable biochemical parameter such as lactate that predicts mortality in many diseases in this scoring system. The investigators named this scoring system HEARTSIL. The investigators aim to compare the diagnostic performance of this score with the diagnostic performance of other scoring systems.

DETAILED DESCRIPTION:
The study was planned to be conducted in Konya City Hospital Emergency Service. Adult patients over 18 years of age who present to the emergency department with chest pain will be included in the study. Patients who do not consent to participate in the study due to chest pain such as ST elevation myocardial infarction, pneumonia, pneumothorax, pulmonary embolism and esophageal rupture will be excluded from the study. Vital signs of the patients, background information, the nature of the pain, the drugs used will be recorded. Blood tests and electrocardiogram will be recorded. Heart Score, TIMI, GRACE score will be calculated. Shock index and lactate value will also be included in the heart score. Shock index 0.5-0.7 = 0 points, 0.71-1 = 1 point and above 1 will be cal-culated as 2 points. Lactate levels 0-2 mEq/L =0 points, between 2,1-3,99 mEq/L= 1 point, above 4 mEq/L levels will be calculated 2 points. These points will be added to the Heart Score and will be named HEARTSIL. Patients will be followed in terms of major cardiac events (MACE) for 3 days and 1 month. Prog-nostic performance of HEARTSIL Score, Heart Score, GRACE, TIMI scores that the investigators developed will be compared.

The data will be uploaded to the database for statistics. First of all, whether the data is normally distributed or not will be determined. Student-t for normally distributed data, Mann-witney-u test for data that are not normally distributed, and chi-square will be used for comparing categorical data. The ROC curve will be drawn and compared in determining the prognostic performance of scoring systems for MACE development. In addition, PPD, NPD, +LR and -LR sensitivity and spe-cificities will be calculated. Values with a p value below 0.05 will be considered statistically signifi-cant.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting to the emergency department with chest pain

Exclusion Criteria:

* ST elevation myocardial infarction,
* Pneumonia, pneumothorax, pulmonary embolism and esophageal rupture
* Patients under 18 years of age
* Pregnant patients
* Patients who do not want to be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chest pain.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-06-14 (Estimated); Study Completion 2021-07-14 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) at 30 days | 30 days after presentation.
  The primary outcome is MACE at 30 days. MACE is a composite outcome of cardiac death, acute myocardial infarction, and coronary revascularization.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) at 3 days | 3 days after presentation.
  The primary outcome is MACE at 3 days. MACE is a composite outcome of cardiac death, acute myocardial infarction, and coronary revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Nazire B Akilli, Assoc Prof, Principal Investigator — Konya City Hospital; Pervin Sagdıc, MD, Study Chair — Konya City Hospital; Turgut Uygun, MD, Study Chair — Konya City Hospital; Ramazan Koylu, Assoc Prof, Study Chair — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No